CLINICAL TRIAL: NCT00435786
Title: Diabetic Patients With End-Stage Renal Disease
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: J.nr. 01 199/02
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2007-02-15 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes; End-Stage Renal Disease; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus; Kidney Failure, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
In diabetic patients with end-stage renal disease to investigate the prevalence of diabetic complications and quality of life and to compare with non-diabetic patients with ESRD and diabetic patients with normal kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Presence of diabetes and treatment with either dialysis or renal transplantation

Exclusion Criteria:

* Age < 18
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke R Sørensen, MD, Principal Investigator — Department of Nephrology, Rigshospitalet